CLINICAL TRIAL: NCT05918549
Title: Movement Analysis in Musculoskeletal Oncology: a Pilot Study
Acronym: AnMov
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Azienda Policlinico Umberto I (Other); Università degli studi di Roma Foro Italico (Other)
Responsible Party: Sponsor
Other Study IDs: RS1704/22
Record Dates: First submitted 2023-03-28; First posted 2023-06-26 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Motion Analysis in Musculoskeletal Oncology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Popolation
  Interventions: Device: Motion Analysis in Musculoskeletal Oncology

INTERVENTIONS:
Device: Motion Analysis in Musculoskeletal Oncology — Noninterventional, prospective, multicenter pilot study of patients with primary and secondary musculoskeletal tumors designed to investigate functional outcomes after therapy using both subjective and quantitative motion detection techniques

SUMMARY:
Noninterventional, prospective, multicenter pilot study of patients with primary and secondary musculoskeletal tumors designed to investigate functional outcomes after therapy using both subjective and quantitative motion detection techniques

ELIGIBILITY:
Inclusion Criteria:

* Age > 6 years
* Diagnosis of primary and secondary tumors of the musculoskeletal system
* Patients who will need to undergo surgery for bone resection or wide excision of soft tissue lesion, and/or radiation or drug treatments
* Availability of follow-up data (for at least 6 months)
* Written informed consent

Exclusion Criteria:

- Inability to perform pre-post treatment assessment

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary and secondary cancers of the musculoskeletal system with estimated survival greater than one year who are candidates for bone resection surgery or wide excision of soft tissue lesion and/or radio and chemotherapy treatments
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-09-28 (Estimated); Study Completion 2024-09-28 (Estimated)

PRIMARY OUTCOMES:
Quality of life | Baseline
  To investigate any differences found using the two methods (quantitative/movement analysis technique versus "subjective"/qualitative technique) in changes in walking/motor characteristics in post-treatment versus pre-treatment.
  Patients will be monitored via a system of wearable sensors (OPAL 15) which send signals to a computer - station receiving. The system is equipped with 15 small, wireless devices and non-invasive, which contain the following sensors:
  i) triaxial accelerometer for measuring linear accelerations of the body segment; ii) triaxial gyroscope for measuring angular speeds; iii) triaxial magnetometer, essential for estimating the orientation of the segment in space corporeal. The system synchronously acquires data from each device and sends it via telemetry to one control unit that collects them and saves them in the local database of the computer used for the acquisition.

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided